CLINICAL TRIAL: NCT01568008
Title: Observational Study of Lumigan® 0.01% for Treatment of Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/GLA/031
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Results first posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-07

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost; Ophthalmic Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Lumigan® 0.01% (bimatoprost 0.01% ophthalmic solution) eye drops at a dose and frequency as determined by the physician.
  Interventions: Drug: Bimatoprost 0.01% ophthalmic solution

INTERVENTIONS:
Drug: Bimatoprost 0.01% ophthalmic solution — Bimatoprost 0.01% ophthalmic solution eye drops at a dose and frequency as determined by the physician.
  Other Names: Lumigan®

SUMMARY:
This is an observational study in patients with POAG or OHT that will collect data on the use of Lumigan® 0.01% (bimatoprost 0.01% ophthalmic solution) in a routine clinical setting. Patients will be seen at baseline and at a follow-up visit approximately 8-12 weeks after baseline, as per normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of POAG or OHT
* Prescribed Lumigan® 0.01%

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with POAG or OHT
Sampling Method: Non-Probability Sample
Enrollment: 933 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Ghent, Oost-Vlaanderen, Belgium

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an observational study of participants who received Lumigan® 0.01% (bimatoprost 0.01% ophthalmic solution) at a dose and frequency as determined by the physician prior to entry into the study.
Period: Overall Study
Arm/Group | All Participants
Started | 933
Completed | 699
Not Completed | 234

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 933
Age Continuous [Mean (Standard Deviation); unit: Years] — Age data was not available for 37 patients.
  Years | 65.40 (11.88)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 442
  Female | 480
  Missing data | 11

OUTCOME MEASURES:

1. Secondary Outcome: Patient Assessment of Treatment Tolerability Using a 4-Point Scale
Description: Patients evaluated their tolerability of treatment using a 4-point scale (very good, good, moderate, and poor). The number of patients assessed in each of the categories is reported.
Time Frame: 12 weeks
Population: All patients with data available for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 888
Participants
  Very good | 460
  Good | 317
  Moderate | 61
  Poor | 50

2. Secondary Outcome: Physician Assessment of Treatment Tolerability Using a 4-Point Scale
Description: The Physician evaluated the patient's tolerability of treatment using a 4-point scale (very good, good, moderate, and poor). The number of patients assessed in each of the categories is reported.
Time Frame: 12 weeks
Population: All patients with data available for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 893
Participants
  Very good | 489
  Good | 331
  Moderate | 49
  Poor | 24

3. Secondary Outcome: Physician Reported Reasons for Treatment Discontinuation
Description: The number of patients who discontinued from treatment by category is reported. More than one reason may apply to each patient.
Time Frame: 12 weeks
Population: All patients with data available for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 87
Participants
  Unacceptable ocular tolerability | 46
  Insufficient IOP control | 20
  Patient lost to follow up | 11
  Patient decision to withdraw from study | 8
  Physician decision to withdraw patient from study | 6
  Other reason | 6

4. Secondary Outcome: Number of Patients Continuing Treatment After 12 Weeks
Description: The number of patients continuing treatment after 12 weeks was determined by the physician answering yes to the question: Is the patient continuing on Lumigan® 0.01% treatment?
Time Frame: 12 weeks
Population: All patients with data available for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 862
Participants | 755

5. Primary Outcome: Intraocular Pressure (IOP) at Baseline
Description: IOP is a measurement of the fluid pressure inside the eye. IOP was measured in the left and right eye at Baseline.
Time Frame: Baseline
Population: All patients with complete data available for IOP.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | All Participants
Number analyzed (Participants) | 889
mm Hg
  Right Eye (n=885) | 22.04 (5.17)
  Left Eye | 22.07 (5.12)

6. Primary Outcome: Intraocular Pressure (IOP) at Week 12
Description: IOP is a measurement of the fluid pressure inside the eye. IOP was measured in the left eye and the right eye at Week 12. The lower the IOP values the greater the improvement.
Time Frame: Week 12
Population: All patients with complete data available for IOP.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | All Participants
Number analyzed (Participants) | 889
mm Hg
  Right Eye (n=885) | 16.94 (3.88)
  Left Eye | 17.02 (4.15)

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 7/933
Other Adverse Events (participants affected / at risk) | 53/933
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=933)
Ocular hyperaemia (Eye disorders) | 3
Vein disorder (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Nightmare (Psychiatric disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=933)
Ocular hyperaemia (Eye disorders) | 53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.